CLINICAL TRIAL: NCT06293872
Title: Evaluation of Two Mini-Implant Lengths in the Infra-Zygomatic Crest Region (A Randomized Clinical Trial, Split-mouth Study)
Brief Title: Evaluation of Two Mini-Implant Lengths in the Infra-Zygomatic Crest Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Abbas Fadhil Alsaeedi, Bachelor's dental Surgery ( B. D. S), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IZC miniscrew
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Orthodontic Appliance Complication
Keywords: mini-screws, infrazygomatic crest zone, IZC, orthodontics implant.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12*2 mm length miniscrew (Experimental): The self-drilling screw is directed at 90° to the occlusal plane at this point. After the initial notch in the bone is created after couple of turns to the driver, the bone screw driver direction is changed by 55°-70° toward the tooth, downward, which aid in bypassing the roots of the teeth and directing the screw to the infra-zygomatic area of the maxilla. The bone screw is screwed until only the head of the screw is visible outside the alveolar mucosa.
  Follow-up: C.B.C.T will be performed after surgery to verify the implant position relative to the adjacent roots.
  Interventions: Device: 12*2 mm length miniscrew
- 14*2 mm length miniscrew (Active Comparator): The self-drilling screw is directed at 90° to the occlusal plane at this point. After the initial notch in the bone is created after couple of turns to the driver, the bone screw driver direction is changed by 55°-70° toward the tooth, downward, which aid in bypassing the roots of the teeth and directing the screw to the infra-zygomatic area of the maxilla. The bone screw is screwed until only the head of the screw is visible outside the alveolar mucosa.
  Follow-up: C.B.C.T will be performed after surgery to verify the implant position relative to the adjacent roots.
  Interventions: Device: 12*2 mm length miniscrew

INTERVENTIONS:
Device: 12*2 mm length miniscrew — Prior to mini-inplant insertion the patient will instructed to rinse mouth with chlorhexidine mouthwash, then local anesthesia will be applied.
  The clinical implication for miniscrew insertion in the IZ crest of adults is 14 to 16 mm above the maxillary occlusal plane and the maxillary first molar.
  The self-drilling screw is directed at 90° to the occlusal plane at this point. After the initial notch in the bone is created after couple of turns to the driver, the bone screw driver direction is changed by 55°-70° toward the tooth, downward, which aid in bypassing the roots of the teeth and directing the screw to the infra-zygomatic area of the maxilla. The bone screw is screwed until only the head of the screw is visible outside the alveolar mucosa.
  Follow-up: C.B.C.T will be performed after surgery to verify the implant position relative to the adjacent roots
  Other Names: 14*2 mm length miniscrew

SUMMARY:
Evaluation of two different lengths of mini-implants in the infrazygomatic area regarding primary stability, pain perception, sinus penetration, secondary stability and failure rate.

DETAILED DESCRIPTION:
orthodontic mini-implants, also known as miniscrew, implants or temporary anchorage devices, offer an effective panacea for Anchorage loss problem during fixed appliance treatments.

Indeed, Mini-implant implantation has become an essential method of controlling anchorage in the clinic and plays an important role in solving some difficult cases, where the integration of orthodontic mini-implants within fixed appliance treatments offers other advantages over conventional anchorage.

Intra-radicular micro-implants are placed in between the roots of teeth (mostly) while extra-radicular bone screws are placed away from the roots in the infra-zygomatic areas (IZC) of the maxilla and the buccal shelf areas (BS) of the mandible. Both extra-radicular bone screws and intra-radicular are classified under temporary anchorage devices used for the purpose of skeletal anchorage.

Due to the limited space, there is a risk of injury to the roots while using Intra-radicular micro-implants. Therefore, the infrazygomatic crest zone is selected as an alternative implantation site in the clinic. The infrazygomatic crest has a double-layered cortex and is close to the maxillary center of the resistance, which is suitable for implantation and provides strong anchorage.

Orthodontic bone screws can be used in almost every clinical situation that a micro-implant is used for, except that they cannot be placed inter-dental purely because of their larger dimension. They can be used for molar uprighting, segmental, and full arch distalization, intrusion of single tooth to full arch, protraction and retraction of dentition and for any other anchorage needs.

the two most specific indications would be - full arch distalization of maxillary and mandibular dentition to camouflage a Class II and a Class III malocclusion and for distalization of arches in re-treatment cases of anchorage loss, which are otherwise difficult to be done with a regular micro-implant or time-consuming.

However, it is adjacent to the maxillary sinus and tooth roots; therefore, we have to consider many factors, such as bone mass, the thickness of the buccal cortex and the relationship with the maxillary sinus and roots, before implantation in the infrazygomatic crest. Furthermore, previous research by our research group found that it is safe to penetrate the maxillary sinus within 1 mm.

This study will be conducted to test the feasibility, reliability of using two different sizes of infrazygomatic mini-implant regarding primary stability, pain perception, sinus penetration, secondary stability, and failure rate.

ELIGIBILITY:
Inclusion Criteria:

- a. Patients (age of patients is 15-50 y.) need metal fixed orthodontic treatment including placement of miniscrews.

b. The position of mini-implant in upper buccal posterior area (infrazygomatic area).

Exclusion Criteria:

* • If c.b.c.t show that the screw placed intraradicular will be excluded.

  * Patient choose to discontinue the treatment was regarded as dropout, since this study pre protocol analysis. exclusion criteria, such as images suggesting
  * Images suggesting sinus inflammation or pathology before mini-implant insertin.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
failure rate | 6 months
  the miniscrew regarded as failed if it is mobile and can not fulfill it is anchorage function, covered by soft tissue.

SECONDARY OUTCOMES:
primary stability | immediately after placement
  primary stability measured for each patient immediately after placemat with use of Dentium stability measuring system (EasyCheck).
secondary stability | after 6months
  secondary stability measured for each patient immediately after placemat with use of Dentium stability measuring system (EasyCheck).
pain perception | after 1st day and after 1st week
  Patients asked to record any pain experienced on the visual analog scale (VAS) score.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi abd Alrubayee, B.D.S; M.Sc; PhD, Study Director — Assistant Professor, Department of Orthodontics, College of Dentistry, University of Baghdad, Iraq.
Locations (1):
- University of Baghdad College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10/10/2024 for 3 months
Access Criteria: I can provide data as word

REFERENCES:
- [Derived] Alsaeedi AF, Alrubayee MA, Sivamurthy G. Evaluation of Two Mini-implant Lengths in the Infrazygomatic Crest Region: A Randomized Clinical Trial. Eur J Dent. 2025 May;19(2):399-408. doi: 10.1055/s-0044-1789015. Epub 2024 Nov 7. PMID 39510519